CLINICAL TRIAL: NCT02849093
Title: Optical Coherence Tomography of Ocular Structures in Epiphora and Dry Eye Syndrome (OCT)
Brief Title: Optical Coherence Tomography of Ocular Structures in Epiphora and Dry Eye Syndrome.
Acronym: OCT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bedford Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 473/2015/387
Record Dates: First submitted 2016-06-17; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Dry Eye Syndrome; Epiphora; Sjögren's Syndrome
Keywords: Optical coherence tomography; imaging of ocular structures
MeSH Terms: conditions — Dry Eye Syndromes; Lacrimal Apparatus Diseases; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Dry Eye Syndrome Patients: Patients who have been diagnosed clinically with Sjögren's will have an OCT image of their lacrimal glands and buccal mucosa taken. Imaging from patients found to have Sjögren's clinically diagnosed following examination of buccal mucosa under the microscope will be compared with images from patients without dry eye syndrome to see of any obvious differences can be identified.
  Interventions: Other: Non-invasive OCT imaging
- Epiphora Patients: Pre and post-operative OCT images of patients undergoing punctoplasty or conjunctivoplasty will be compared to images of the same structures in people without watery eyes.
  Interventions: Other: Non-invasive OCT imaging
- Asymptomatic Patients: OCT images will be captured of the cornea, conjunctiva, lacrimal gland and buccal mucosa to establish normal appearance in asymptomatic patients.
  Interventions: Other: Non-invasive OCT imaging

INTERVENTIONS:
Other: Non-invasive OCT imaging — Optical Coherence Tomography (OCT) to capture high resolution cross-sectional images of tissue microstructures using infra-red radiation.

SUMMARY:
The primary aim of the study is to investigate whether optical coherence tomography (OCT) may be a useful tool for investigating the in-vivo histology of ocular structures in patients with tear film pathology. In epiphora the investigators will image the proximal lacrimal system. In dry eye syndrome the investigators will image the lacrimal gland and also the buccal mucosa.

The secondary aim of the study is to investigate the appearance of the normal cornea and conjunctiva under OCT imaging.

DETAILED DESCRIPTION:
Optical Coherence Tomography (OCT) is a safe and non-invasive method of high resolution cross-sectional imaging of tissue microstructures using infra-red radiation. It was first described by Huang et al in 1991.

The principle of OCT imaging is similar to ultrasound; infra-red light is shone at a tissue of interest and the reflectivity of each layer within the tissue gives rise to a signal that enables a cross-sectional picture of the tissue to be constructed. In contrast to ultrasound however, it is not possible to use the timing of reflected pulses of light to infer the distance of the reflecting surface. This is because of the extremely high velocity of light (3x10^8 ms^-1), which would require the detector to have a temporal resolution of a few tens of femtoseconds in order to provide a spatial resolution of 10 microns within the tissue under observation. therefore, interferometry is applied to the infra-red light source in order to determine the distance that reflected light has travelled.

OCT currently has a wide range of applications including imaging the retina, the anterior chamber of the eye and the endothelium of the coronary arteries (when used intravascularly). It has also been used in preclinical cancer research to image tumours. IT has a resolution of 1-20µm and can penetrate approximately 1-2mm into tissue.

Dry Eye Syndrome:

Sjögren's is a common cause of dry eye syndrome. Currently a biopsy of the lacrimal gland is required to establish the diagnosis. In this study the investigators explore whether it is possible to distinguish the lacrimal gland in Sjögren's patients from the normal lacrimal gland using OCT imaging. The investigators will also image the buccal mucosa of suspected Sjögren's patients and compare the results to previously published images of the normal mucosa.

Epiphora:

Punctal anatomy is clinically relevant in the management of epiphora because punctal stenosis is one of the many causes of this condition. However, there are currently no routinely used imaging modalities or objective quantitative assessment systems for the proximal lacrimal system.

OCT seems to be ideally suited to imaging the punctum due to its high resolution and non-invasive nature. The investigators have recently completed a study demonstrating the feasibility of OCT imaging of the proximal lacrimal system in a cohort of subjects with normal ocular anatomy and no symptoms of epiphora. In this study the investigators will examine the practical clinical applications of OCT imaging pre and post-operatively in patients undergoing punctoplasty or conjunctivoplasty to treat epiphora.

Asymptomatic Patients:

The investigators aim to establish the normal OCT appearance of the conjunctiva and cornea; and also aim to establish the normal appearance of the lacrimal gland and the buccal mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Patients with watery eyes who are listed for punctoplasty surgery
* Patients with dry eyes secondary to Sjögren's (i.e. presence of anti-Ro/SSA or La/SSB autoantibodies, reduced Schirmer's test less than 5mm over 5 minutes without local anaesthesia or typical clinical presentation).
* Members of staff at our eye clinic with no history of previous ocular surgery or watering/dryness.

Exclusion Criteria:

* Previous eyelid or lacrimal surgery
* Patients without capacity to consent
* Patients unwilling to participate
* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmology Patients (dry eye syndrome & epiphora), Inflammatory and Immune System Patients, asymptomatic subjects
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Qualitative difference in OCT appearance of lacrimal and buccal glands measured at a single time-point, between dry eye patients and asymptomatic patients | Baseline, at the time of listing for surgery
  OCT images of the lacrimal gland and buccal mucosa will be taken from dry eye patients and asymptomatic patients. These images will be compared qualitatively, to determine if there are any differences in the appearance of the lacrimal and buccal glands under OCT, in patients with dry eye disease compared to healthy subjects.
Comparison of punctual diameter, canalicular diameter and canalicular depth between asymptomatic patients and patients with epiphora pre-operatively and post-operatively, and correlation with Lac-Q questionnaire score | 26 weeks
  All patients with epiphora who are due to undergo punctoplasty (for punctual stenosis) or conjunctivoplasty (for conjunctivochalasis) will have pre- and post-operative imaging of their left and right lower punctum / conjunctiva respectively. Patients will also have their epiphora symptoms graded according to the Lac Q questionnaire before and after surgery. Asymptomatic patients will have OCT imaging taken of the cornea and conjunctiva.

CONTACTS AND LOCATIONS:
Overall Officials: Anant Sharma, FRCOphth, Principal Investigator — Moorfields at Bedford